CLINICAL TRIAL: NCT04133402
Title: Evaluation of Fertility of Patients With a History of Postpartum Hemorrhage, Complicating Low-dose Delivery With Intrauterine Tamponade Treatment
Brief Title: Fertility After Intrauterine Tamponing Balloon: Where Are we
Acronym: FERTIBTIU
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_89; 2018-A01609-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2019-10

CONDITIONS: Hemorrhage Postpartum; Fertility Disorders
Keywords: Hemorrhage Post-partum; Fertility; Uterine balloon tamponade; Vaginal Birth
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today, few data are available on the patient's fertility following intrauterine tamponade balloon (BTIU) used for postpartum hemorrhage (PPH) after vaginal delivery (AVB). Several studies have concluded that there are no fertility disorders after conservative surgical treatment or embolization. BTIU is an essential treatment in the management of PPH. The aim was to evaluate post-BTIU fertility and the appearance of gynecological symptoms.

This is a bicentric retrospective study (Valenciennes, Lille, France), between 2012 and 2017. The data will be collected by telephone interview on fertility and various gynecological functional symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal birth
* Post partum haemorrhage
* Intrauterine tamponing balloon
* Between 2012 and 2017
* CHRU Lille and CH Valenciennes

Exclusion Criteria:

* Minor patients
* Initial intake started in another center (postpartum transfer).
* Refusal to participate in the study
* Invasive treatments for postpartum haemorrhage
* Caesarean

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients with postpartum haemorrhage after vaginal delivery between 2012 and 2017 in Valenciennes maternity and the CHRU Lille, treated by intrauterine tamponade therapy.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Frequency of infertility | 7 years
  defined as the absence of pregnancy after 12 months of attempted pregnancy.

SECONDARY OUTCOMES:
Time to obtain a new pregnancy evaluating the stop of contraceptionand desire for pregnancy | 7 years
Frequency of gynecological complications after use of an intrauterine tamponade balloon. | 7 years
Type of gynecological complications after use of an intrauterine tamponade balloon. | 7 years
  type = infections , pelvic pain, cycle disorders
the frequency of obstetric complications for the next pregnancy | 7 years
type of obstetrical complications | 7 years
  complications = intrauterine growth retardation, threat of premature labor
Frequency of recurrent postpartum haemorrhage in the next pregnancy | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Garabedian, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France